CLINICAL TRIAL: NCT06349005
Title: Hemodynamic Response to Various Laryngoscopes During Tracheal Intubation in CABG Patients
Brief Title: Laryngoscopy and Coronary Artery Bypass Graft Surgery
Acronym: VL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Prof. Dr, Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111
Record Dates: First submitted 2024-02-26; First posted 2024-04-05 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Videolaryngoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group Storz VL (Active Comparator): Patients will undergo intubation with the Storz Videolaryngoscope®, during which their hemodynamic responses will be documented.
  Interventions: Other: Tracheal intubation using Storz VL
- Group MacGrath VL (Active Comparator): Patients will undergo intubation with the McGrath Videolaryngoscope®, during which their hemodynamic responses will be documented.
  Interventions: Other: Tracheal intubation using MacGrath VL
- Group EzVision VL (Active Comparator): Patients will undergo intubation with the EzVision Videolaryngoscope®, during which their hemodynamic responses will be documented.
  Interventions: Other: Tracheal intubation using EzVision VL
- Group Traditional (Active Comparator): Patients will undergo intubation with the traditional (Macintosh) laryngoscopy, during which their hemodynamic responses will be documented.
  Interventions: Other: Tracheal intubation using Macintosh laryngoscopy

INTERVENTIONS:
Other: Tracheal intubation using Storz VL — Video-assisted intubation technique using Storz VL
  Arms: Group Storz VL
Other: Tracheal intubation using Macintosh laryngoscopy — Traditional intubation technique using Macintosh laryngoscopy
  Arms: Group Traditional
Other: Tracheal intubation using MacGrath VL — Video-assisted intubation technique using MacGrath VL
  Arms: Group MacGrath VL
Other: Tracheal intubation using EzVision VL — Video-assisted intubation technique using EzVision VL
  Arms: Group EzVision VL

SUMMARY:
In this prospective, randomized, controlled trial, the purpose is to compare Macintosh laryngoscope, EzVision® video laryngoscope, McGrath® video laryngoscope and Storz® video laryngoscope in terms of hemodynamic response associated with intubation in adult patients undergoing Coronary Artery Bypass Surgery (CABG).

DETAILED DESCRIPTION:
During endotracheal intubation, laryngoscopy can significantly affect hemodynamic responses, including tachycardia and elevated blood pressure, which may be particularly detrimental to individuals with cardiovascular conditions. Various studies have explored the hemodynamic reactions associated with laryngeal stimulation through different intubation devices. Researchers hypothesize that endotracheal intubation using video laryngoscopy will elicit a reduced hemodynamic response compared to traditional (Macintosh) laryngoscopy. In this prospective and randomized clinical study, the purpose is to compare the Macintosh laryngoscope, EzVision® video laryngoscope, McGrath® video laryngoscope and Storz® video laryngoscope concerning haemodynamic response associated with intubation in adult patients undergoing Coronary Artery Bypass Surgery (CABG).

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18 and 75 years.
* Scheduled for elective coronary artery bypass surgery.
* Classified under American Society of Anesthesiologists (ASA) physical status II-III.
* Patients with no history of difficult intubation or associated risk factors.

Exclusion Criteria:

* Emergency case
* Predicted difficult airways
* Body mass index > 35 kilograms per meter squared
* Baseline hemodynamic instability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2025-01-12 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Hemodynamic response | Change from baseline Systolic or Diastolic or mean Blood Pressure at 10 minutes
  Change from baseline invasive blood pressure
Hemodynamic response | Change from baseline heart rate at 10 minutes
  Change from baseline heart rate

SECONDARY OUTCOMES:
Intubation time | 180 seconds
  The duration from when the laryngoscope passes through the teeth until it is withdrawn back to the teeth will be measured.
Visualization of the glottis | 180 seconds
  According to Cormack Lehane classification four grades (1-4). The higher the grade, the higher the likelihood of difficult intubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)